CLINICAL TRIAL: NCT02377258
Title: IBD Cancer and Serious Infection in Europe
Acronym: I-CARE
Status: Completed | Type: Observational
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Other Study IDs: GETAID 2015-01
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: IBD
Keywords: Lymphoma; safety; biologic therapies
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- 1: without previous or ongoing exposure to IS or biologics, (5ASA and Steroids are allowed)
  Interventions: Other: Non Interventional
- 2: with on-going anti-TNF monotherapy
  Interventions: Other: Non Interventional
- 3: with thiopurines monotherapy
  Interventions: Other: Non Interventional
- 4: with on-going combination therapy
  Interventions: Other: Non Interventional
- 5: patients on vedolizumab (1 on vedolizumab alone and 1 on combination therapy)
  Interventions: Other: Non Interventional
- 6: patients on ustekinumab (alone or on combination therapy)
  Interventions: Other: Non Interventional

INTERVENTIONS:
Other: Non Interventional

SUMMARY:
The primary objective of I-CARE is to assess prospectively the presence and the extent of safety concerns (cancers, especially, lymphoma, and serious infections risks) for anti-TNF alone or in combination with thiopurines among IBD patients.

We will stratify the risk of cancers and serious infections according to IBD phenotype and disease activity (clinical, radiologic and endoscopic).

DETAILED DESCRIPTION:
The four main secondary objectives of the I-CARE project are:

* To investigate prospectively the impact of anti-TNF based strategies on the natural history of IBD and their potential for disease modification by collecting validated surrogate markers such as mucosal healing and disease complications such as bowel damage (strictures, fistulas, abscess), surgeries, and hospitalizations
* To assess the evolution of Patient Reported Outcome (ePRO) on a yearly basis and the impact of anti-TNF agents on ePRO in IBD
* To evaluate the benefit-risk ratio of strategies based on an earlier and wider use of anti-TNF therapy for IBD
* To assess the healthcare costs and cost-efficacy of current therapeutic strategies in IBD 5-ASA and Steroids across Europe At least 5000 IBD patients treated with 5-ASA or Steroids and FU for 3 years

  * use of 5-ASA and efficacy (persistence, switch, mucosal healing etc.)
  * chemoprevention of CRC: first study that will specifically and accurately address this question
  * use of budesonide mmx and efficacy (clinical efficacy, mucosal healing and potential for disease modification)
  * safety of steroids (infections etc)

STUDY DESIGN:

22 patients per investigator. Each Investigator will recruit and enrol 20 patients with imposed treatment stratification : Group 1: 5 without previous or ongoing exposure to IS or biologics, (5 ASA and Steroids are allowed) Group 2: 5 with on-going anti-TNF monotherapy Group 3: 5 with thiopurines monotherapy Group 4: 5 with on-going combination therapy Group 5: 2 patients on vedolizumab (on vedolizumab alone and 1 on combination therapy) (optionnal) Group 6: 5 patients treated with ustekinumab with or without any concomitant medications. (optional)

ELIGIBILITY:
Inclusion Criteria:

* CD or UC
* Capable to complete eDiary on a regular basis, and have access to smartphone or internet
* Accepted to participate and provide personal information (name, phone and email) for contact
* Accepted to be contacted by study coordinators on a regular basis for follow up with missing information

Exclusion Criteria:

* Unable to sign consent
* Unable to access internet or use smartphone
* Refused to sign consent or to provide personal identification information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 17600 patients in 17 European countries, enrolled by 800 investigators (22 subjects per investigator)
Sampling Method: Non-Probability Sample
Enrollment: 13262 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
assess prospectively the presence and the extent of safety concerns (cancers, especially, lymphoma, and serious infections risks) for anti-TNF alone or in combination with thiopurines among IBD patients. | 3 years
  assess prospectively the presence and the extent of safety concerns (cancers, especially, lymphoma, and serious infections risks) for anti-TNF alone or in combination with thiopurines among IBD patients.

SECONDARY OUTCOMES:
Disease modification | 3 Years
  To investigate prospectively the impact of anti-TNF based strategies on the natural history of IBD and their potential for disease modification by collecting validated surrogate markers such as mucosal healing and disease complications such as bowel damage (strictures, fistulas, abscess), surgeries, and hospitalisations
ePRO | 3 Years
  To assess the evolution of Patient Reported Outcome (ePRO) on a yearly basis and the impact of anti-TNF agents on ePRO in IBD
Benefit-Risk | 3 Years
  To evaluate the benefit-risk ratio of strategies based on an earlier and wider use of anti-TNF therapy for IBD
Cost Efficacy | 3 Years
  To assess the healthcare costs and cost-efficacy of current therapeutic strategies in IBD

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Peyrin-Biroulet, MD, PhD, Principal Investigator — Head of IBD Unit Inserm U954 Nancy University Hospital FRANCE
Locations (1):
- Chu Nancy, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Peyrin-Biroulet L, Nazar M, Sheahan A, Geldhof A, Azzabi A, Baert F, Mailhat C, Rousseau H, Rahier JF, Beaugerie L. Long-term safety of ustekinumab in Crohn's disease: Descriptive analysis from an observational post-authorisation safety study using I-CARE cohort data. Dig Liver Dis. 2026 Jan;58(1):74-81. doi: 10.1016/j.dld.2025.09.026. Epub 2025 Oct 25. PMID 41139534
- [Derived] Peyrin-Biroulet L, Rahier JF, Kirchgesner J, Abitbol V, Shaji S, Armuzzi A, Karmiris K, Gisbert JP, Bossuyt P, Helwig U, Burisch J, Yanai H, Doherty GA, Magro F, Molnar T, Lowenberg M, Halfvarson J, Zagorowicz E, Rousseau H, Baumann C, Baert F, Beaugerie L; I-CARE Collaborator Group. I-CARE, a European Prospective Cohort Study Assessing Safety and Effectiveness of Biologics in Inflammatory Bowel Disease. Clin Gastroenterol Hepatol. 2023 Mar;21(3):771-788.e10. doi: 10.1016/j.cgh.2022.09.018. Epub 2022 Sep 22. PMID 36152897